CLINICAL TRIAL: NCT00881556
Title: A Pilot Study of Reduced Intensity Conditioning (RIC) and Allogeneic Stem Cell Transplantation (ALLOSCT) In Children With Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: Allogeneic Stem Cell Transplantation (ALLOSCT) in Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Acronym: RDEB
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD5420; CHNY-08-536 (Other: CUMC)
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Epidermolysis Bullosa
Keywords: Allogeneic Stem Cell Transplant; AlloSCT; RDEB; recessive dystrophic epidermolysis bullosa
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica | interventions — Fibroblast Growth Factor 7; fludarabine; fludarabine phosphate; Busulfan; Lorazepam; Alemtuzumab; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RIC Group (Experimental): Reduced Intensity Transplant Conditioning (RIC):
  Palifermin (Kepivance®) 60 mcg/kg/day for 6 days Fludarabine 30 mg/m2 IV x 1 for 6 days Busulfan 4 mg/kg/day IV divided BID for 4 days Lorazepam 0.02-0.05 mg/kg for 5 days Alemtuzumab 20 mg/m2 IV for 5 days Tacrolimus 0.03mg/kg/24 hours as continuous infusion for 4 days
  Interventions: Drug: Palifermin; Drug: Fludarabine; Drug: Busulfan; Drug: Lorazepam; Drug: Alemtuzumab; Drug: Tacrolimus

INTERVENTIONS:
Drug: Palifermin — 60 mcg/kg/day for 6 days
  Other Names: Kepivance
Drug: Fludarabine — 30 mg/m2 IV x 1 for 6 days
  Other Names: Fludara
Drug: Busulfan — 4 mg/kg/day IV divided BID for 4 days
  Other Names: Myleran
Drug: Lorazepam — 0.02-0.05 mg/kg for 5 days
  Other Names: Ativan
Drug: Alemtuzumab — 20 mg/m2 IV for 5 days
  Other Names: Lemtrada
Drug: Tacrolimus — 0.03mg/kg/24 hours as continuous infusion for 4 days
  Other Names: Prograf; Protopic; Hecoria

SUMMARY:
Reduced Intensity Conditioning (RIC) and Allogeneic Stem Cell Transplantation (AlloSCT) from family-related donors and unrelated cord blood (UCB) donors will be safe and well tolerated in selected patients with RDEB.

To determine the event-free survival (EFS) and overall survival (OS) following RIC consisting of busulfan/fludarabine/alemtuzumab (BFA) and AlloSCT in selected patients with RDEB.

DETAILED DESCRIPTION:
Epidermolysis bullosa (EB), is a diverse group of genodermatoses, which is considered a rare and orphan disease and affects approximately 1 in 20,000 people in the United States for a cumulative total of close to 20,000[1-4]. There are three major subtypes of inherited EB, including EB simplex (EBS), junctional EB (JEB), and dystrophic EB[1-4]. RDEB is among the most severe and represents approximately 10% of all forms of EB[1-4]. A rough estimate would then project that there are several thousand patients with RDEB in the U.S. at the current time. Up to 30 different clinical phenotypes and mutations in at least 10 structural genes in different sub-types of EB have been reported[4-8]. In addition to heritable subtypes of EB, there is an acquired autoimmune form in which the patients develop auto-antibodies directed against similar proteins of the inherited dystrophic forms of EB, including EB acquisita (EBA).

We have previously reported our experience with RIC with BFA [48] in pediatric AlloSCT recipients (mean age 9.5 yrs [1.4-21], 11/4 M/F, 10 non-malignant, 5 malignant disease, [6 sibling, 5 UCB, 5 matched unrelated donor]); median time to ANC ≥ 500/mm3 and platelet count ≥20K/mm3 was 22 and 30 days, respectively. Probability of day +180 and 365 donor chimerism was 90% (Figure 7), and OS was 95% (Figure 8). This conditioning regimen therefore results in a high degree of donor chimerism and survival with minimal regimen related mortality.

ELIGIBILITY:
Inclusion Criteria:

* Recessive Dystrophic Epidermolysis Bullosa (RDEB)
* Diagnosis of RDEB using molecular diagnosis and sequencing of mutations
* Skin biopsy to determine status of type VII collagen
* Age ≤21 years
* Patient must have adequate organ function as below:

  1. Adequate renal function defined as:

     * Serum creatinine less than or equal to 1.5 x normal, or
     * Creatinine clearance or radioisotope glomerular filtration rate (GFR) =40 ml/min/m2 or > 60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range
  2. Adequate liver function defined as:

     * Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase (AST)) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase (ALT))< 5.0 x normal
  3. Adequate cardiac function defined as:

     * Shortening fraction of ≥28% by echocardiogram, or
     * Ejection fraction of ≥48% by radionuclide angiogram or echocardiogram
  4. Adequate pulmonary function defined as:

     * Uncorrected diffusing capacity of the lungs for carbon monoxide (DLCO) ≥35% by pulmonary function test
     * For children who are uncooperative, no evidence of dyspnea at rest

Exclusion Criteria:

* Karnofsky/Lansky Performance Score <50%
* Pregnant or nursing
* Uncontrolled bacterial, viral or mold infection
* History or presence of skin squamous cell carcinoma

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2009-08-20 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 2 years
Overall Survival (OS) | Up to 2 years

SECONDARY OUTCOMES:
Percentage of whole blood (CD45), T-cell (CD3), and NK cell (CD56) chimerism following RIC and AlloSCT in selected patients with RDEB | Up to Day +730
Percentage of donor skin dermal chimerism following RIC and AlloSCT in selected patients with RDEB. | Up to Day +730

CONTACTS AND LOCATIONS:
Overall Officials: Angela Christiano, PhD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - The Children's Hospital, Aurora, Colorado
  - Children's Memorial Hospital, Chicago, Illinois
  - Morgan Stanley Children's Hospital of NYP, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided